CLINICAL TRIAL: NCT06950840
Title: Intravenous Dipyrone Compared With Intravenous Acetaminophen for Maternal Fever During Labor: A Randomised Controlled Trial
Brief Title: Antipyretic Treatment for Intrapartum Fever: Dipyrone vs Acetaminophen (RCT)
Acronym: PARADIP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, ilia kleiner, Specialist Obstetrician & Gynecologist; Director of Labor-and-Delivery Rooms and the Maternity Department, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WOMC-0093-25
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Intrapartum Fever; Chorioamnionitis
Keywords: maternal fever; labour; acetaminophen; dipyrone; metamizole
MeSH Terms: conditions — Chorioamnionitis | interventions — Acetaminophen; Dipyrone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dipyrone (Experimental): Dipyrone IV 1 g once
  Interventions: Drug: dipyrone
- Acetaminophen (Experimental): Acetaminophen 1 g IV once
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 1 g IV once
  Arms: Acetaminophen
Drug: dipyrone — Dipyrone IV 1 g once
  Arms: Dipyrone

SUMMARY:
Chorioamnionitis, or intraamniotic infection, is a common condition affecting 2-5% of all term births. This condition poses well-recognized maternal and neonatal risks, and entails a series of clinical management decisions concerning both the mother and neonate. Therefore, timely detection and treatment of chorioamnionitis is of paramount importance. The occurrence of chorioamnionitis is associated with a higher risk of labor abnormalities, which increase the risk of cesarean delivery (CD) 3 to 4 fold.

As recommended by current guidelines, treatment of suspected intraamniotic infection should include broad-spectrum antibiotics. In addition, the use of antipyretics is advocated. This is particularly important during the intrapartum period since fetal acidosis in the setting of fever has been associated with a marked increase in the incidence of neonatal encephalopathy. Maternal fever even in the absence of documented fetal acidosis is associated with adverse neonatal outcomes, particularly neonatal encephalopathy, though it is unclear to what extent the etiology of the fever rather than the fever itself is causative . Furthermore, treating intrapartum fever with antipyretics may also be helpful in reducing fetal tachycardia thereby avoiding the tendency to perform cesarean for a non-reassuring fetal status. Nevertheless, it remains understudied which is the most appropriate antipyretic agent in this regard, where both dipyrone and acetaminophen are safe alternatives . Antipyretic agent with a faster onset of action may be preferable in this setting.

DETAILED DESCRIPTION:
Chorioamnionitis, or intraamniotic infection, affects 2-5% of term deliveries and is associated with significant maternal and neonatal risks, including a 3- to 4-fold increase in cesarean delivery. Management includes prompt antibiotic treatment and antipyretic use, particularly during labor, where maternal fever may contribute to fetal acidosis and increased risk of neonatal encephalopathy. Even in the absence of acidosis, maternal fever alone is linked to adverse neonatal outcomes. Antipyretics may also help resolve fetal tachycardia, potentially avoiding unnecessary cesarean sections. While both dipyrone and acetaminophen are considered safe, it remains unclear which has superior efficacy in the intrapartum setting, and an agent with faster onset may offer clinical advantages.

Stages of study: Following the diagnosis of suspected intrapartum intraamniotic infection, eligible women will be offered to participate. All women will be treated with the same broad-spectrum antibiotic regimen. As stated above, those who gave their informed consent will be randomly assigned to either dipyrone or acetaminophen.

After administering antipyretic treatment, oral temperature will be monitored every 5 minutes for up to 40 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a trial of vaginal delivery, with suspected intra-amniotic infection defined as isolated maternal fever of 39°C or greater, or an sustained oral temperature of 38-38.9°C for at least 30 minutes or with one or more of the following: maternal leukocytosis, purulent cervical drainage, or fetal tachycardia.

Exclusion Criteria:

* Known history of adverse events for dipyrone or acetaminophen
* Age <18 years
* Gestational age <24 weeks
* Intrauterine fetal death
* Fever onset prior to delivery
* Known liver disease
* Known leukopenia
* In addition, those who will develop allergic event or any adverse event possible related to any of the antipyretics used will be excluded from the

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified women who are pregnant and meet inclusion criteria for suspected intra-amniotic infection during labor.
Enrollment: 140 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Time to defervesce | 120 min
  Time (minutes) from drug administration to temperature < 38 °C

SECONDARY OUTCOMES:
Time to resolution of fetal tachycardia | 120 min
  Time to resolution of fetal tachycardia (min)
Mode of delivery | From enrollment to delivery
  Mode of delivery (vaginal / cesarean)
Apgar scores | At 1 and 5 minutes after birth
  Apgar scores - Standard newborn assessment
Neonatal arterial pH level | Immediately after birth
  Neonatal arterial pH level

CONTACTS AND LOCATIONS:
Overall Officials: Ilia Kleiner, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
Time to defervescence, fetal heart rate response, delivery mode, Apgar scores, neonatal pH
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months after study completion; available for 2 years
Access Criteria: Qualified researchers with institutional ethics approval will be able to access de-identified individual participant data, including time to fever resolution, fetal heart rate response, delivery mode, Apgar scores, and neonatal arterial pH. Data will be available upon reasonable request to the Principal Investigator via email. Requests must include a brief study proposal and evidence of ethical approval. If approved, data will be shared in a secure, password-protected format. Supporting documents such as the study protocol and statistical analysis plan will also be made available upon request.